CLINICAL TRIAL: NCT07073430
Title: Research on the Application Evaluation of Artificial Intelligence Supported System in Assisting the Diagnosis of Colorectal Tubular Adenoma Lesions
Brief Title: Evaluation of Artificial Intelligence System in Diagnosis of Colorectal Tubular Adenoma Lesions
Status: Recruiting | Type: Observational
Sponsor: Renmin Hospital of Wuhan University (Other)
Collaborators: Beijing Friendship Hospital, Captial Medical University (Unknown); Air Force Military Medical University, China (Other); The Sixth Affiliated Hospital, Sun Yat-sen University (Unknown); Army Medical University, China (Other); Guizhou Provincial People's Hospital (Other); Shengjing Hospital (Other); Zhejiang University (Other); Shandong University (Other); The Second Medical Center of The General Hospital of the People's Liberation Army (Unknown)
Responsible Party: Principal Investigator, ChenMingkai, Professor, Wuhan University
Other Study IDs: WDRY2024-K153
Record Dates: First submitted 2025-07-09; First posted 2025-07-18 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-06

CONDITIONS: Colorectal Adenoma; Artificial Intelligence (AI) in Diagnosis
Keywords: Colorectal Adenoma; Artificial Intelligence (AI) in Diagnosis
MeSH Terms: interventions — Narrow Band Imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Traditional colonoscopy examination group: the system shows the original colonoscopy video.
- AI-assisted colonoscopy examination group: the system presents the detected polyp location with a hollow blue alert box directly on a high definition monitor,marking whether it is an adenoma or not and the probability of it.
  Interventions: Device: AI models with NBI

INTERVENTIONS:
Device: AI models with NBI — AI models for detecting intestinal adenoma in magnifying endoscopy with NBI.
  Groups: AI-assisted colonoscopy examination group

SUMMARY:
This study is a prospective,multi-center and observational clinical study.Investigators would like to innovatively construct a "trinity" database of colorectal tubular adenomas based on white light - magnifying chromo - pathological images.It simulates the decision - making logic of doctors, and based on the multimodal endoscopic LAFEQ method previously proposed, develop a multimodal deep - learning diagnostic model for colon adenomas and an interpretable risk prediction model for intestinal adenomas. While achieving high - precision auxiliary treatment decisions, clearly present the decision - making basis, and break through the limitation of poor interpretability of previous medical imaging AI models.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥ 18 years, who need to undergo colonoscopy, regardless of gender.
* Voluntarily sign the informed consent form
* Promise to abide by the research procedures and cooperate in the implementation of the entire research process.

Exclusion Criteria:

* Patients who has a history of abdominal or pelvic surgery or radiotherapy in the past;
* Patients who has definite active lower gastrointestinal bleeding.
* Existing or suspected hereditary colorectal polyposis, inflammatory bowel disease;
* Uncontrolled hypertension (systolic blood pressure > 160 mmHg or diastolic blood pressure > 95 mmHg after standardized treatment)
* There is a history of stroke, coronary artery disease, or vascular disease;
* Pregnant;
* Intestinal preparation cannot be carried out.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who need to undergo colonoscopy are enrolled in this study.
Sampling Method: Non-Probability Sample
Enrollment: 4200 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2026-10-31 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
The accuracy rate of diagnosing adenomas | during endoscopy
  The accuracy rate of the endoscopic AI model in diagnosing adenomas (presence or absence of adenomas, number of adenomas, advanced adenomas).

SECONDARY OUTCOMES:
The prediction for the disease risk level | during endoscopy
  The prediction rate of the interpretable artificial intelligence-assisted diagnosis model for the disease risk level.

CONTACTS AND LOCATIONS:
Overall Officials: Mingkai Chen, PHD, Principal Investigator — Renmin Hospital of Wuhan University
Locations (1):
- Renmin Hospital of Wuhan University, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Strum WB. Colorectal Adenomas. N Engl J Med. 2016 Mar 17;374(11):1065-75. doi: 10.1056/NEJMra1513581. No abstract available. PMID 26981936
- [Background] Glissen Brown JR, Mansour NM, Wang P, Chuchuca MA, Minchenberg SB, Chandnani M, Liu L, Gross SA, Sengupta N, Berzin TM. Deep Learning Computer-aided Polyp Detection Reduces Adenoma Miss Rate: A United States Multi-center Randomized Tandem Colonoscopy Study (CADeT-CS Trial). Clin Gastroenterol Hepatol. 2022 Jul;20(7):1499-1507.e4. doi: 10.1016/j.cgh.2021.09.009. Epub 2021 Sep 14. PMID 34530161
- [Background] Yao L, Li X, Wu Z, Wang J, Luo C, Chen B, Luo R, Zhang L, Zhang C, Tan X, Lu Z, Zhu C, Huang Y, Tan T, Liu Z, Li Y, Li S, Yu H. Effect of artificial intelligence on novice-performed colonoscopy: a multicenter randomized controlled tandem study. Gastrointest Endosc. 2024 Jan;99(1):91-99.e9. doi: 10.1016/j.gie.2023.07.044. Epub 2023 Aug 1. PMID 37536635
- [Background] Wallace MB, Sharma P, Bhandari P, East J, Antonelli G, Lorenzetti R, Vieth M, Speranza I, Spadaccini M, Desai M, Lukens FJ, Babameto G, Batista D, Singh D, Palmer W, Ramirez F, Palmer R, Lunsford T, Ruff K, Bird-Liebermann E, Ciofoaia V, Arndtz S, Cangemi D, Puddick K, Derfus G, Johal AS, Barawi M, Longo L, Moro L, Repici A, Hassan C. Impact of Artificial Intelligence on Miss Rate of Colorectal Neoplasia. Gastroenterology. 2022 Jul;163(1):295-304.e5. doi: 10.1053/j.gastro.2022.03.007. Epub 2022 Mar 15. PMID 35304117
- [Background] Haight TJ, Eshaghi A. Deep Learning Algorithms for Brain Imaging: From Black Box to Clinical Toolbox? Neurology. 2023 Mar 21;100(12):549-550. doi: 10.1212/WNL.0000000000206808. Epub 2023 Jan 13. No abstract available. PMID 36639238
- [Background] Stahlschmidt SR, Ulfenborg B, Synnergren J. Multimodal deep learning for biomedical data fusion: a review. Brief Bioinform. 2022 Mar 10;23(2):bbab569. doi: 10.1093/bib/bbab569. PMID 35089332
- [Background] van der Velden BHM, Kuijf HJ, Gilhuijs KGA, Viergever MA. Explainable artificial intelligence (XAI) in deep learning-based medical image analysis. Med Image Anal. 2022 Jul;79:102470. doi: 10.1016/j.media.2022.102470. Epub 2022 May 4. PMID 35576821
- [Background] Wang Y, Zhen L, Tan TE, Fu H, Feng Y, Wang Z, Xu X, Goh RSM, Ng Y, Calhoun C, Tan GSW, Sun JK, Liu Y, Ting DSW. Geometric Correspondence-Based Multimodal Learning for Ophthalmic Image Analysis. IEEE Trans Med Imaging. 2024 May;43(5):1945-1957. doi: 10.1109/TMI.2024.3352602. Epub 2024 May 2. PMID 38206778
- [Background] Tempany CM, Jayender J, Kapur T, Bueno R, Golby A, Agar N, Jolesz FA. Multimodal imaging for improved diagnosis and treatment of cancers. Cancer. 2015 Mar 15;121(6):817-27. doi: 10.1002/cncr.29012. Epub 2014 Sep 9. PMID 25204551
- [Background] Zhou T, Cheng Q, Lu H, Li Q, Zhang X, Qiu S. Deep learning methods for medical image fusion: A review. Comput Biol Med. 2023 Jun;160:106959. doi: 10.1016/j.compbiomed.2023.106959. Epub 2023 Apr 20. PMID 37141652
- [Background] Dekker E, Rex DK. Advances in CRC Prevention: Screening and Surveillance. Gastroenterology. 2018 May;154(7):1970-1984. doi: 10.1053/j.gastro.2018.01.069. Epub 2018 Feb 15. PMID 29454795
- [Background] Li J, Zhu Y, Dong Z, He X, Xu M, Liu J, Zhang M, Tao X, Du H, Chen D, Huang L, Shang R, Zhang L, Luo R, Zhou W, Deng Y, Huang X, Li Y, Chen B, Gong R, Zhang C, Li X, Wu L, Yu H. Development and validation of a feature extraction-based logical anthropomorphic diagnostic system for early gastric cancer: A case-control study. EClinicalMedicine. 2022 Mar 30;46:101366. doi: 10.1016/j.eclinm.2022.101366. eCollection 2022 Apr. PMID 35521066